CLINICAL TRIAL: NCT01031511
Title: A Randomised Controlled Trial on the Effect of Cognitive-behavioural Therapy for High-functioning Children With Autistic Spectrum Disorder
Brief Title: Effect of Cognitive Behavioural Therapy (CBT) for Children With Autistic Spectrum Disorders
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Healthcare Group, Singapore (Other Government)
Collaborators: Nanyang Technological University (Other); Autism Resource Centre, Singapore (Unknown)
Responsible Party: Min, Sung / Dr., Institute of Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DSRB Ref Code: A/05/091; NMRC/1002/2005 (Other Grant/Funding Number: National Medical Research Council (Singapore)); 130/2005 (Other: Institute of Mental Health (Singapore) Clinical Research Committee)
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Last update posted 2009-12-14 (Estimated); Status verified 2009-02

CONDITIONS: Autism Spectrum Disorder; Anxiety
Keywords: High-Functioning Autistic Spectrum Disorder; Anxiety; Cognitive Behavioural Therapy; Social Recreational; Parent Stress
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group - CBT (Experimental)
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Control Group (No Intervention)
  Interventions: Other: Social Recreational

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — 16 weekly sessions of 1.5 hrs in small groups of 3-4 children conducted by 2 therapists
  Arms: Treatment Group - CBT
Other: Social Recreational — 16 weekly sessions of 1.5 hrs in small groups of 3-4 children, conducted by 2 therapists
  Arms: Control Group

SUMMARY:
Cognitive Behavioural Therapy is an effective intervention program for children with High-Functioning Autistic Spectrum Disorder to remediate anxiety issues.

ELIGIBILITY:
Inclusion Criteria:

* Assessed to have Autistic Spectrum Disorder, Asperger Syndrome, Pervasive Developmental Disorder, Not Otherwise Specified by the DSM-IV criteria, based on clinical interview, Asperger Syndrome Diagnostic Scale (ASDS) or Autism Diagnostic Observation Schedule (ADOS)
* Child have a Verbal Comprehension Index of 80 and Perceptual Reasoning Index of 90 and above
* No change of medication dosage 1 month prior to the commencement of program for the child and through out the duration of the study
* Written parental consent and assent from children above 12 years old

Exclusion Criteria:

* Children with Verbal Comprehension Index of 80 and Perceptual Reasoning Index of 90 and below.
* Children who are undergoing other Cognitive Behavioural treatment program concurrently
* Those without parental consent will not be able to participate

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2005-06; Primary Completion 2010-01 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Anxiety level of child | Pre Treatment, Post-treatment, 3 months follow-up, 6 months follow-up, One year follow-up

SECONDARY OUTCOMES:
Parent Stress Level | Pre Treatment, Post-treatment, 3 months follow-up, 6 months follow-up, One year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Min Sung, Principal Investigator — Institute of Mental Health, Singapore
Locations (1):
- Institute of Mental Health, Singapore, Singapore, Singapore